CLINICAL TRIAL: NCT02465138
Title: A Randomized Controlled Trial of IV Ketorolac to Prevent Post-ERCP Pancreatitis
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Lack of Funding
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 15-16365
Record Dates: First submitted 2015-03-25; First posted 2015-06-08 (Estimated); Last update posted 2022-04-28 (Actual); Status verified 2022-04

CONDITIONS: Pancreatitis
MeSH Terms: conditions — Pancreatitis | interventions — Ketorolac; Ketorolac Tromethamine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Placebo (Placebo Comparator): Normal Saline will be administered prior to procedure.
  Interventions: Drug: Placebo
- Toradol (Active Comparator): Intravenous ketorolac prior to ERCP
  Interventions: Drug: Ketorolac

INTERVENTIONS:
Drug: Ketorolac — Intravenous ketorolac
  Other Names: Toradol
  Arms: Toradol
Drug: Placebo — Intravenous saline
  Arms: Placebo

SUMMARY:
Determine if IV ketorolac is an effective agent in the prevention of post-ERCP pancreatitis. Determine if IV ketorolac provides improved post-procedure analgesia.

Determine if systemic mediators of inflammation are reduced in patients receiving IV ketorolac following ERCP.

DETAILED DESCRIPTION:
Acute pancreatitis is the most common major complication of both diagnostic and therapeutic endoscopic retrograde cholangiopancreatography (ERCP), accounting for substantial morbidity and an annual expenditure of approximately 150 million annually.(1,2) Non-steroidal anti-inflammatory agents (NSAIDs) have been shown to be effective in multiple prospective randomized controlled trial for the prevention of post-ERCP pancreatitis.(3-6) NSAIDs are postulated to inhibit phospholipase A2 and prostaglandin synthesis, which plays an important role in the inflammatory cascade in acute pancreatitis. Rectal suppository indomethacin (a potent COX-2 inhibitor) has been effective in preventing post-ERCP pancreatitis in clinical trials and is now recommended for routine use for ERCP by the European Society of Gastrointestinal Endoscopy.(7) Toradol® (ketorolac), an NSAID available in IV form, is a more potent COX-2 inhibitor and analgesic than indomethacin.(8,9) Ketorolac is routinely used postoperatively following major surgery to assist in pain control particularly following orthopedic procedures. IV ketorolac has never been evaluated for the prevention of post-ERCP pancreatitis.

ELIGIBILITY:
Inclusion Criteria:

* All patients presenting to SFGH for ERCP
* Age 18-85
* Do not meet exclusion criteria

Exclusion Criteria:

* Acute pancreatitis at the time of ERCP
* Use of NSAIDs in the previous week
* Peptic ulcer disease
* Severe renal dysfunction
* Pregnancy
* Lithium therapy
* allergy to ketorolac

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-11 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events | 5 days after ERCP procedure

CONTACTS AND LOCATIONS:
Overall Officials: John P Cello, MD, Principal Investigator — University of California, San Francisco
Locations (2):
- United States (2):
  - San Francisco General Hospital, San Francisco, California
  - UCSF/San Francisco General Hospital, San Francisco, California

REFERENCES:
- [Background] Freeman ML, Guda NM. Prevention of post-ERCP pancreatitis: a comprehensive review. Gastrointest Endosc. 2004 Jun;59(7):845-64. doi: 10.1016/s0016-5107(04)00353-0. No abstract available. PMID 15173799
- [Background] Freeman ML, Nelson DB, Sherman S, Haber GB, Herman ME, Dorsher PJ, Moore JP, Fennerty MB, Ryan ME, Shaw MJ, Lande JD, Pheley AM. Complications of endoscopic biliary sphincterotomy. N Engl J Med. 1996 Sep 26;335(13):909-18. doi: 10.1056/NEJM199609263351301. PMID 8782497
- [Background] Elmunzer BJ, Scheiman JM, Lehman GA, Chak A, Mosler P, Higgins PD, Hayward RA, Romagnuolo J, Elta GH, Sherman S, Waljee AK, Repaka A, Atkinson MR, Cote GA, Kwon RS, McHenry L, Piraka CR, Wamsteker EJ, Watkins JL, Korsnes SJ, Schmidt SE, Turner SM, Nicholson S, Fogel EL; U.S. Cooperative for Outcomes Research in Endoscopy (USCORE). A randomized trial of rectal indomethacin to prevent post-ERCP pancreatitis. N Engl J Med. 2012 Apr 12;366(15):1414-22. doi: 10.1056/NEJMoa1111103. PMID 22494121
- [Background] Otsuka T, Kawazoe S, Nakashita S, Kamachi S, Oeda S, Sumida C, Akiyama T, Ario K, Fujimoto M, Tabuchi M, Noda T. Low-dose rectal diclofenac for prevention of post-endoscopic retrograde cholangiopancreatography pancreatitis: a randomized controlled trial. J Gastroenterol. 2012 Aug;47(8):912-7. doi: 10.1007/s00535-012-0554-7. Epub 2012 Feb 18. PMID 22350703
- [Background] Sotoudehmanesh R, Khatibian M, Kolahdoozan S, Ainechi S, Malboosbaf R, Nouraie M. Indomethacin may reduce the incidence and severity of acute pancreatitis after ERCP. Am J Gastroenterol. 2007 May;102(5):978-83. doi: 10.1111/j.1572-0241.2007.01165.x. Epub 2007 Mar 13. PMID 17355281
- [Background] Khoshbaten M, Khorram H, Madad L, Ehsani Ardakani MJ, Farzin H, Zali MR. Role of diclofenac in reducing post-endoscopic retrograde cholangiopancreatography pancreatitis. J Gastroenterol Hepatol. 2008 Jul;23(7 Pt 2):e11-6. doi: 10.1111/j.1440-1746.2007.05096.x. Epub 2007 Aug 7. PMID 17683501
- [Background] Dumonceau JM, Andriulli A, Deviere J, Mariani A, Rigaux J, Baron TH, Testoni PA; European Society of Gastrointestinal Endoscopy. European Society of Gastrointestinal Endoscopy (ESGE) Guideline: prophylaxis of post-ERCP pancreatitis. Endoscopy. 2010 Jun;42(6):503-15. doi: 10.1055/s-0029-1244208. Epub 2010 May 26. PMID 20506068
- [Background] Cryer B, Feldman M. Cyclooxygenase-1 and cyclooxygenase-2 selectivity of widely used nonsteroidal anti-inflammatory drugs. Am J Med. 1998 May;104(5):413-21. doi: 10.1016/s0002-9343(98)00091-6. PMID 9626023
- [Background] Gillis JC, Brogden RN. Ketorolac. A reappraisal of its pharmacodynamic and pharmacokinetic properties and therapeutic use in pain management. Drugs. 1997 Jan;53(1):139-88. doi: 10.2165/00003495-199753010-00012. PMID 9010653
- [Background] Gross V, Leser HG, Heinisch A, Scholmerich J. Inflammatory mediators and cytokines--new aspects of the pathophysiology and assessment of severity of acute pancreatitis? Hepatogastroenterology. 1993 Dec;40(6):522-30. PMID 7509768
- [Background] Bhatia M, Brady M, Shokuhi S, Christmas S, Neoptolemos JP, Slavin J. Inflammatory mediators in acute pancreatitis. J Pathol. 2000 Feb;190(2):117-25. doi: 10.1002/(SICI)1096-9896(200002)190:23.0.CO;2-K. PMID 10657008
- [Background] Makela A, Kuusi T, Schroder T. Inhibition of serum phospholipase-A2 in acute pancreatitis by pharmacological agents in vitro. Scand J Clin Lab Invest. 1997 Aug;57(5):401-7. doi: 10.3109/00365519709084587. PMID 9279965
- [Background] Murray B, Carter R, Imrie C, Evans S, O'Suilleabhain C. Diclofenac reduces the incidence of acute pancreatitis after endoscopic retrograde cholangiopancreatography. Gastroenterology. 2003 Jun;124(7):1786-91. doi: 10.1016/s0016-5085(03)00384-6. PMID 12806612
- [Background] Cheon YK, Cho KB, Watkins JL, McHenry L, Fogel EL, Sherman S, Schmidt S, Lazzell-Pannell L, Lehman GA. Efficacy of diclofenac in the prevention of post-ERCP pancreatitis in predominantly high-risk patients: a randomized double-blind prospective trial. Gastrointest Endosc. 2007 Dec;66(6):1126-32. doi: 10.1016/j.gie.2007.04.012. PMID 18061712
- [Background] Senol A, Saritas U, Demirkan H. Efficacy of intramuscular diclofenac and fluid replacement in prevention of post-ERCP pancreatitis. World J Gastroenterol. 2009 Aug 28;15(32):3999-4004. doi: 10.3748/wjg.15.3999. PMID 19705494
- [Background] Dobronte Z, Toldy E, Mark L, Sarang K, Lakner L. [Effects of rectal indomethacin in the prevention of post-ERCP acute pancreatitis]. Orv Hetil. 2012 Jun 24;153(25):990-6. doi: 10.1556/OH.2012.29403. Hungarian. PMID 22714033
- [Background] Helleberg L. Clinical Pharmacokinetics of indomethacin. Clin Pharmacokinet. 1981 Jul-Aug;6(4):245-58. doi: 10.2165/00003088-198106040-00001. PMID 7249487